CLINICAL TRIAL: NCT05717023
Title: Online Guided Self-help Intervention for Sexual Distress Following Sexual Assault: A Single Case Experimental Study
Brief Title: Guided Self-help Following Sexual Assault - SCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Holloway University (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Kimberley Khoo, Principal Investigator, Trainee Clinical Psychologist, Royal Holloway University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3379
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Sexual Assault; Sexual Dysfunction; Sex Disorder
Keywords: sexual distress
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Single case experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online guided self-help intervention for sexual distress following sexual assault (Experimental): The intervention only has one arm. All participants will be provided 4 sessions of guided self-help intervention to be completed once weekly.
  Interventions: Behavioral: Online guided self-help intervention for sexual distress following sexual assault

INTERVENTIONS:
Behavioral: Online guided self-help intervention for sexual distress following sexual assault — 4 Sessions of guided self-help will be shared with the participants. These will be in the form of handout and video recordings that participant access through Qualtrics. The intervention is based on research on sexual trauma, psychosexual difficulties and materials developed by Bart's NHS Foundation Trust Sexual Wellbeing Service. It has been made in collaboration with clinicians within the service, experts by experience and the chief investigator.Within the document there are scripts for each session which are read out in the video recordings. The handouts depict the visual images for the video and the materials provided to participant.

SUMMARY:
This single-case experimental design aims to evaluate the acceptability & feasibility of an online guided self-help intervention for female survivors of sexual assault who experience difficulties returning to sex.

The main questions it aims to answer are:

• Is the intervention viewed as acceptable by female survivors of sexual assault? Acceptability is defined as as how willing participants are to use the materials and their satisfaction with its content.

The secondary question is, are there initial indicators that the intervention is effective? Effectiveness is measured by a reduction in the measure of sexual distress and improvement of sexual satisfaction - specifically confidence and motivation in practising strategies that will improve their experience of sex.

Participants will complete the intervention independently. There will be 4-sessions which involve watching videos, with one session completed weekly. The developed materials aim to to help women understand their difficulties, learn practical strategies and build confidence in returning to sex. The materials are also guided by a piloted group for sexual distress by Bart's National Health Service (NHS) trust Sexual Wellbeing Service. The NHS is the publicly funded healthcare system in England.

DETAILED DESCRIPTION:
The study adopts a non-concurrent AB single-case experimental design (SCED) with follow-up. Although AB designs are not sufficient to test treatment effectiveness, using this study type informs the feasibility of the intervention. In addition, a multiple baseline approach was adopted where participants will be randomly allocated to different lengths of baselines ranging from 5 to 14 days in Phase A. Phase B consists of a 4- week intervention period where participants complete idiographic measures daily. Follow-up will be completed one month after the intervention.

Potential participants will complete an online screening questionnaire via Qualtrics. Eligible participants who provide consent will complete the baseline questionnaires such as the Female Sexual Function Index, Female Sexual Distress Scale and State Self Compassion Scale. Afterwards, participants will be randomly allocated to different baseline lengths (5 to 14 days) for Phase A.

Participants complete visual analogue scales daily for the length of Phase A. Following Phase A, participants begin Phase B, completing the intervention weekly for four weeks. Visual analogue scales are completed daily during phase B.

Follow-up occurs four weeks after Phase B. Participants complete the Female Sexual Function Index, Female Sexual Distress Scale, State Self Compassion Scale, Client Satisfaction Questionnaire and a qualitative feedback form.

ELIGIBILITY:
Inclusion Criteria:

* Cis female
* Experience of sexual assault (in adulthood or childhood but not within the previous 12 months)
* Experiencing sexual distress/difficulties
* United Kingdom Resident
* Willingness to complete guided self help
* Aged 18 and above
* Ability to read and understand English to provide informed consent and meaningfully engage with the self-help materials
* Ability to access online guided self-help material through a computer or phone

Exclusion Criteria:

* experiencing severe acute mental health difficulties
* sexual assault occurring within the last 12 months
* currently experiencing more than fleeting suicidal thoughts or engaging in severe self-harming (individuals who have been sexually assaulted are likely to experience suicidal thoughts or self harm behaviours, individuals with fleeting suicidal thoughts or superficial self harm with strong protective factors may be included however, since there is no contact with mental health professionals during the intervention unless participants reach out for triage, it is difficult to assess risk and participants have to be excluded if they do not have social support systems of are currently accessing psychological support).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis female
Enrollment: 20 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | At follow up, 8 weeks
  The client satisfaction questionnaire is an 8-item questionnaire scored on a 4-point scale and will be provided to participants at follow up to ask the acceptability and satisfaction towards the intervention. Permission has been asked to adapt the questionnaire to focus on satisfaction for the intervention instead of service satisfaction. Total scores range from 8 to 32 with higher scores indicating higher satisfaction.
Feedback Form | At follow up, 8 weeks
  A short qualitative feedback form will be provided to participants. This form has been developed with experts by experience and will have open ended questions for participants to provide more detailed feedback about the intervention. The questionnaire is only used at follow up.

SECONDARY OUTCOMES:
Baseline Visual Analogue Scales | Completed daily up to 2 weeks
  Visual analogue scales are scales with two ends. Participants will be asked to rate on the line how much they agree or disagree with a statement. Visual analogue scales are used to measure the following concepts: shame, guilt, self-criticism, compassion, normalising and motivation. The scales were developed for this research project in collaboration with experts by experience.
Intervention Visual Analogue Scales | Completed daily up to 1 month
  Visual analogue scales are scales with two ends. Participants will be asked to rate on the line how much they agree or disagree with a statement. Visual analogue scales are used to measure the following concepts: shame, guilt, self-criticism, compassion, normalising and motivation. The scales were developed for this research project in collaboration with experts by experience.
Female Sexual Distress scale - Revised (FSDS-R) | Baseline and 8 weeks
  The Female Sexual Distress Scale - Revised is used to assess distress related to sex in women. This 13-item self-report questionnaire is scored has five points, (0: never; 1: rarely; 2: occasionally; 3: frequently; 4: always). Total scores range from 0 to 52 with higher scores indicating higher levels of sexual distress.
Female Sexual Function Index (FSFI) | Baseline and 8 weeks
  The Female Sexual Function Index is a 19-item questionnaire that measures six domains: desire, arousal, lubrication, orgasm, satisfaction and pain. The questionnaire uses a 5-point likert scale and is scored from 1 to 5. Total score range from 2 to 36 with lower scores indicating higher levels of difficulties.
State Self Compassion Questionnaire (SSCS-S) | Baseline and 8 weeks
  The State Self Compassion Questionnaire is a 6-item questionnaire scored on a 5-point scale from 1 (not very true for me) to 5 (very true for me). The scale was not develop to indicate high or low levels of state self-compassion rather it is to be used in a comparative manner to examine the change in compassion after the intervention. The minimum score is 1 and the maximum score is 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Vosper, Principal Investigator — Bart's NHS Foundation Trust
Locations (1):
- Bart's Sexual Wellbeing Service, National Health Service, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: research protocol (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05717023/Prot_SAP_000.pdf
  • Study Protocol: intervention manual (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT05717023/Prot_001.pdf